CLINICAL TRIAL: NCT00002963
Title: Cutaneous Absorption and Intralesional Penetration of Topical Amino-Levulinic Acid in Basal Cell Carcinoma and Squamous Cell Carcinoma as Measured by In Situ Fluorescence and Intensified Video Fluorescence Microscopy
Brief Title: Photodynamic Therapy in Treating Patients With Skin Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: DS 92-42; RPCI-DS-92-42; NCI-V97-1191
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2013-01

CONDITIONS: Non-melanomatous Skin Cancer
Keywords: basal cell carcinoma of the skin; squamous cell carcinoma of the skin
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — Aminolevulinic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: aminolevulinic acid hydrochloride
Procedure: conventional surgery

SUMMARY:
RATIONALE: Photodynamic therapy uses light and drugs that make cancer cells more sensitive to light to kill tumor cells. Photodynamic therapy using aminolevulinic acid cream may be effective in treating patients with skin cancer.

PURPOSE: This randomized phase II trial is studying how well photodynamic therapy works in treating patients with skin cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Characterize the penetration of topically applied aminolevulinic acid (ALA) into the lesions of patients with primary basal cell and squamous cell carcinomas.
* Quantitate the depth of fluorescence achievable with varying application periods of ALA in these patients.
* Compare the results of tissue fluorescence with surface fluorescence measurements in these patients.

OUTLINE: This is a randomized study. Patients are stratified according to lesion type (superficial basal cell carcinoma (BCC) vs nodular BCC vs squamous cell carcinoma). Patients within each group are randomized to receive one of two application times: 4-5 or 20-24 hours in duration.

Aminolevulinic acid is topically applied either in a cream mixture or an alcohol base and an occlusive dressing placed over the lesion. After the randomized treatment duration has expired, the dressing is removed and quantitative protoporphyrin IX fluorescence measurements from the tumor and surrounding skin are mapped using a fluorometer. Routine surgical excision is then performed on the carcinoma.

Patients return after one to two weeks for a follow-up examination and suture removal.

PROJECTED ACCRUAL: 54 patients will be accrued within 10 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven basal cell carcinoma or squamous cell carcinoma
* Candidate for complete surgical excision

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* No inflammation or infection of treated area

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Biopsy at least 2 weeks prior to surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1993-11; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Depth of penetration of aminolevulinic acid as measured by the accumulation of protoporphyrin IX

CONTACTS AND LOCATIONS:
Overall Officials: Allan R. Oseroff, MD, PhD, Study Chair — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States